CLINICAL TRIAL: NCT06980259
Title: Spatially Fractionated Radiotherapy Versus Conventional Radiotherapy in the Treatment of Soft Tissue Sarcoma:A Multicenter，Prospective, Phase II, Randomized Controlled Trial
Brief Title: Spatially Fractionated Radiotherapy Versus Conventional Radiotherapy in the Treatment of Soft Tissue Sarcoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinbo Yue, Director of Department Radiation Oncology, Shandong Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDZLEC2025-075-02
Record Dates: First submitted 2025-05-12; First posted 2025-05-20 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-04

CONDITIONS: Soft Tissue Sarcoma (STS)
Keywords: Soft Tissue Sarcoma; Spatially Fractionated Radiotherapy; Objective Response Rate; Conventional Radiotherapy
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Intervention Model Description: This multicenter, prospective, randomized phase II trial compares the efficacy and safety of Spatially Fractionated Radiation Therapy (SFRT) vs. Conventional Radiation Therapy (CRT) in soft tissue sarcoma (STS, tumor diameter ≥5 cm). 106 patients are randomized 1:1. CRT delivers 3.0 Gy/fraction for 15-20 fractions using IMRT or IMPT. SFRT adds weekly high-dose vertices (8-15 Gy/fraction, 3-4 fractions) to CRT, using IMRT, IMPT, or VMAT to create a grid-like dose pattern. Both groups use IGRT for precise target volume (GTV, CTV, PTV) definition. Primary endpoint is ORR at 3, 6, 9, and 12 months post-radiotherapy (RECIST 1.1/Choi criteria). Secondary endpoints include 1-year LC, PFS, safety (CTCAE v5.0), and QoL (EORTC QLQ-C30).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spatially Fractionated Radiotherapy (SFRT) Group (Experimental): SFRT builds on CRT, administered at 3.0 Gy per fraction for 15-20 fractions, with the addition of weekly high-dose vertices of 8-15 Gy per fraction for 3-4 fractions. It utilizes Intensity-Modulated Radiation Therapy (IMRT), Intensity-Modulated Proton Therapy (IMPT), or Volumetric Modulated Arc Therapy (VMAT) to create a grid-like pattern of alternating high- and low-dose regions.
  Interventions: Radiation: Spatially Fractionated Radiotherapy
- Conventional Radiotherapy (CRT) Group (Active Comparator): CRT is delivered at 3.0 Gy per fraction for a total of 15-20 fractions, utilizing Intensity-Modulated Radiation Therapy (IMRT) or Intensity-Modulated Proton Therapy (IMPT) techniques, ensuring a target volume dose coverage of at least 90%.
  Interventions: Radiation: Conventional Radiotherapy

INTERVENTIONS:
Radiation: Spatially Fractionated Radiotherapy — SFRT builds on CRT, administered at 3.0 Gy per fraction for 15-20 fractions, with the addition of weekly high-dose vertices of 8-15 Gy per fraction for 3-4 fractions. It employs Intensity-Modulated Radiation Therapy (IMRT), Intensity-Modulated Proton Therapy (IMPT), or Volumetric Modulated Arc Therapy (VMAT) to create a grid-like pattern of alternating high- and low-dose regions. Target volume delineation includes the gross tumor volume (GTV), clinical target volume (CTV, expanded 0.5-1.0 cm from GTV), and planning target volume (PTV, expanded 1.0 cm from CTV). Prior to each treatment session, cone-beam CT (CBCT) or kilovoltage cone-beam CT (kV-CBCT) is used for Image-Guided Radiation Therapy (IGRT) to verify patient positioning.
  Arms: Spatially Fractionated Radiotherapy (SFRT) Group
Radiation: Conventional Radiotherapy — CRT is delivered at 3.0 Gy per fraction for a total of 15-20 fractions, utilizing Intensity-Modulated Radiation Therapy (IMRT) or Intensity-Modulated Proton Therapy (IMPT) techniques, ensuring a target volume dose coverage of at least 90%. Target volume delineation includes the gross tumor volume (GTV), clinical target volume (CTV, expanded 0.5-1.0 cm from GTV), and planning target volume (PTV, expanded 1.0 cm from CTV). Prior to each treatment session, cone-beam CT (CBCT) or kilovoltage cone-beam CT (kV-CBCT) is used for Image-Guided Radiation Therapy (IGRT) to verify patient positioning.
  Arms: Conventional Radiotherapy (CRT) Group

SUMMARY:
This study is a multicenter, prospective, randomized controlled phase II clinical trial designed to evaluate the efficacy and safety of Spatially Fractionated Radiation Therapy (SFRT) compared to Conventional Radiation Therapy (CRT) in the treatment of soft tissue sarcoma (STS, minimum tumor diameter ≥5 cm). A total of 106 patients were enrolled and randomized in a 1:1 ratio. The primary endpoint is the objective response rate (ORR) of the target lesion at 3, 6, 9, and 12 months post-radiotherapy, assessed using RECIST 1.1 and Choi criteria. Secondary endpoints include the 1-year local control rate (LC) of the target lesion, progression-free survival (PFS), safety (per CTCAE v5.0), and quality of life (QoL, assessed by EORTC QLQ-C30). CRT is delivered at 3.0 Gy per fraction for a total of 15-20 fractions. SFRT comprises CRT at 3.0 Gy per fraction for 15-20 fractions, augmented by weekly high-dose vertices of 8-15 Gy per fraction for 3-4 fractions, aiming to enhance tumor control and potentially stimulate immune responses.

This study is a multicenter, prospective, randomized controlled phase II clinical trial designed to evaluate the efficacy and safety of Spatially Fractionated Radiation Therapy (SFRT) compared to Conventional Radiation Therapy (CRT) in the treatment of soft tissue sarcoma (STS, minimum tumor diameter ≥5 cm). A total of 106 patients were enrolled and randomized in a 1:1 ratio. The primary endpoint is the objective response rate (ORR) of the target lesion at 3, 6, 9, and 12 months post-radiotherapy, assessed using RECIST 1.1 and Choi criteria. Secondary endpoints include the 1-year local control rate (LC) of the target lesion, progression-free survival (PFS), safety (per CTCAE v5.0). CRT is delivered at 3.0 Gy per fraction for a total of 15-20 fractions. SFRT comprises CRT at 3.0 Gy per fraction for 15-20 fractions, augmented by weekly high-dose vertices of 8-15 Gy per fraction for 3-4 fractions, aiming to enhance tumor control and potentially stimulate immune responses.

DETAILED DESCRIPTION:
This study is a multicenter, prospective, randomized controlled phase II clinical trial designed to systematically compare the efficacy and safety of Spatially Fractionated Radiation Therapy (SFRT) versus Conventional Radiation Therapy (CRT) in the treatment of soft tissue sarcoma (STS, minimum tumor diameter ≥5 cm). STS is a malignant tumor with low radiosensitivity, and CRT yields limited objective response rates (ORR) and local control rates (LC). The study employs Intensity-Modulated Radiation Therapy (IMRT), Intensity-Modulated Proton Therapy (IMPT), or Volumetric Modulated Arc Therapy (VMAT) techniques. CRT is administered at 3.0 Gy per fraction for a total of 15-20 fractions. SFRT builds on CRT at 3.0 Gy per fraction for 15-20 fractions, supplemented by weekly high-dose vertices of 8-15 Gy per fraction for 3-4 fractions, aiming to enhance tumor control and stimulate potential immune responses.

A total of 106 patients will be enrolled and randomized 1:1 into the SFRT and CRT arms (53 patients per arm). The primary endpoint is the ORR of the target lesion at 3, 6, 9, and 12 months post-radiotherapy, assessed using RECIST 1.1 and Choi criteria. Secondary endpoints include the 1-year LC of the target lesion, progression-free survival (PFS), safety (per CTCAE v5.0).

Eligibility criteria include patients aged 18-70 years, ECOG performance status ≤2, and an expected survival of ≥3 months, excluding those with secondary primary tumors or severe organ dysfunction. Comprehensive baseline assessments (imaging, pathology, and laboratory tests) are conducted before treatment. Toxicity is monitored weekly during treatment, with ≥grade 3 toxicities prompting treatment suspension. Efficacy evaluations are performed at 3, 6, 9, and 12 months post-radiotherapy, with follow-up scheduled every 3 months in the first year, every 6 months in the second year, and annually thereafter. Statistical analysis is based on a one-sided α=0.05 and β=0.8, anticipating an ORR of 40% for SFRT compared to 15% for CRT.

Through its multicenter design and rigorous evaluation, this study aims to validate whether SFRT can improve ORR in STS, providing scientific evidence to optimize radiotherapy strategies, enhance patient prognosis, and improve QoL. Additionally, it seeks to offer insights into the treatment of other radioresistant tumors.

This study is a multicenter, prospective, randomized controlled phase II clinical trial designed to systematically compare the efficacy and safety of Spatially Fractionated Radiation Therapy (SFRT) versus Conventional Radiation Therapy (CRT) in the treatment of soft tissue sarcoma (STS, minimum tumor diameter ≥5 cm). STS is a malignant tumor with low radiosensitivity, and CRT yields limited objective response rates (ORR) and local control rates (LC). The study employs Intensity-Modulated Radiation Therapy (IMRT), Intensity-Modulated Proton Therapy (IMPT), or Volumetric Modulated Arc Therapy (VMAT) techniques. CRT is administered at 3.0 Gy per fraction for a total of 15-20 fractions. SFRT builds on CRT at 3.0 Gy per fraction for 15-20 fractions, supplemented by weekly high-dose vertices of 8-15 Gy per fraction for 3-4 fractions, aiming to enhance tumor control and stimulate potential immune responses.

A total of 106 patients will be enrolled and randomized 1:1 into the SFRT and CRT arms (53 patients per arm). The primary endpoint is the ORR of the target lesion at 3, 6, 9, and 12 months post-radiotherapy, assessed using RECIST 1.1 and Choi criteria. Secondary endpoints include the 1-year LC of the target lesion, progression-free survival (PFS), safety (per CTCAE v5.0).

Eligibility criteria include patients aged 18-70 years, ECOG performance status ≤2, and an expected survival of ≥3 months, excluding those with secondary primary tumors or severe organ dysfunction. Comprehensive baseline assessments (imaging, pathology, and laboratory tests) are conducted before treatment. Toxicity is monitored weekly during treatment, with ≥grade 3 toxicities prompting treatment suspension. Efficacy evaluations are performed at 3, 6, 9, and 12 months post-radiotherapy, with follow-up scheduled every 3 months in the first year, every 6 months in the second year, and annually thereafter. Statistical analysis is based on a one-sided α=0.05 and β=0.8, anticipating an ORR of 40% for SFRT compared to 15% for CRT.

Through its multicenter design and rigorous evaluation, this study aims to validate whether SFRT can improve ORR in STS, providing scientific evidence to optimize radiotherapy strategies, enhance patient prognosis, and improve QoL. Additionally, it seeks to offer insights into the treatment of other radioresistant tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18-70 years, irrespective of gender. 2. Pathologically or clinically confirmed diagnosis of soft tissue sarcoma. 3. Minimum tumor diameter ≥5 cm. 4. Receiving systemic treatment as per multidisciplinary team (MDT) recommendations.

  5. Measurable lesion (per RECIST 1.1/Choi criteria: longest diameter >1.5 cm, or >1 cm with two measurable perpendicular diameters).

  6. ECOG performance status ≤2. 7. Expected survival ≥3 months. 8. Normal liver, kidney, lung, and cardiac function, with tolerance for treatment.

  9. Patients of childbearing potential agree to use reliable contraception during treatment and for one year thereafter.

  10. Voluntary provision of signed informed consent.

Exclusion Criteria:

* (1) Patients with a second primary malignancy. (2) Diagnosis of aggressive fibromatosis or rhabdomyosarcoma. (3) Prior radiotherapy to the target lesion. (4) Tumor unsuitable for radiotherapy. (5) Severe liver, kidney, lung, or cardiac dysfunction, precluding tolerance to systemic therapy or radiotherapy.

  (6) Other severe medical conditions that may impact the study (e.g., uncontrolled diabetes, gastric ulcers, or other serious cardiopulmonary diseases).

  (7) Severe or uncontrolled infections, or active autoimmune diseases. (8) Clinically evident central nervous system dysfunction. (9) Pregnant or lactating women, or women of childbearing potential not using contraception.

  (10) Other conditions deemed unsuitable for participation by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2027-05-20 (Estimated); Study Completion 2028-05-20 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 3、6、9、12months
  The objective response rate (ORR) is defined as the proportion of patients with soft tissue sarcoma target lesions achieving complete response (CR) or partial response (PR) at 3, 6, 9, and 12 months post-radiotherapy, evaluated according to RECIST 1.1 and Choi criteria. Per RECIST 1.1, CR is defined as the complete disappearance of all target lesions, and PR is defined as a ≥30% reduction in the sum of the diameters of target lesions. Per Choi criteria, CR is defined as the complete disappearance of all target lesions, and PR is defined as a ≥10% reduction in the sum of the diameters of target lesions or a ≥15% decrease in tumor density (Hounsfield Units, HU) on CT scans.

SECONDARY OUTCOMES:
Safety Assessment | 1 year
  Adverse events (e.g., skin reactions, tissue fibrosis, organ dysfunction) are monitored during treatment and follow-up in accordance with the CTCAE v5.0 criteria.
Local Control Rate（LC) | 1year
  The local control rate (LC) is defined as the proportion of patients with no progression of the radiotherapy target lesion (i.e., no local recurrence or tumor enlargement, evaluated according to RECIST 1.1 criteria) one year after radiotherapy.
Progression-Free Survival （PFS) | 1 year
  Progression-free survival (PFS) is defined as the time from the start of radiotherapy to either progression of the target lesion (assessed per RECIST 1.1 criteria) or patient death from any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Jinbo Yue, Doctor, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu P, Wang S, Zhou J, Yuan K, Wang X, Li L, Lang J, Lu S. Spatially fractionated radiotherapy (Lattice SFRT) in the palliative treatment of locally advanced bulky unresectable head and neck cancer. Clin Transl Radiat Oncol. 2024 Jul 30;48:100830. doi: 10.1016/j.ctro.2024.100830. eCollection 2024 Sep. PMID 39219705
- [Background] Moghaddasi L, Reid P, Bezak E, Marcu LG. Radiobiological and Treatment-Related Aspects of Spatially Fractionated Radiotherapy. Int J Mol Sci. 2022 Mar 20;23(6):3366. doi: 10.3390/ijms23063366. PMID 35328787
- [Background] Billena C, Khan AJ. A Current Review of Spatial Fractionation: Back to the Future? Int J Radiat Oncol Biol Phys. 2019 May 1;104(1):177-187. doi: 10.1016/j.ijrobp.2019.01.073. Epub 2019 Jan 23. PMID 30684666
- [Background] Yang JC, Chang AE, Baker AR, Sindelar WF, Danforth DN, Topalian SL, DeLaney T, Glatstein E, Steinberg SM, Merino MJ, Rosenberg SA. Randomized prospective study of the benefit of adjuvant radiation therapy in the treatment of soft tissue sarcomas of the extremity. J Clin Oncol. 1998 Jan;16(1):197-203. doi: 10.1200/JCO.1998.16.1.197. PMID 9440743
- [Background] Siegel RL, Miller KD, Jemal A. Cancer statistics, 2020. CA Cancer J Clin. 2020 Jan;70(1):7-30. doi: 10.3322/caac.21590. Epub 2020 Jan 8. PMID 31912902
- [Background] Yan W, Khan MK, Wu X, Simone CB 2nd, Fan J, Gressen E, Zhang X, Limoli CL, Bahig H, Tubin S, Mourad WF. Spatially fractionated radiation therapy: History, present and the future. Clin Transl Radiat Oncol. 2019 Oct 22;20:30-38. doi: 10.1016/j.ctro.2019.10.004. eCollection 2020 Jan. No abstract available. PMID 31768424
- [Background] Owen D, Harmsen WS, Ahmed SK, Petersen IA, Haddock MG, Ma DJ, Pulsipher S, Corbin KS, Lester SC, Park SS, Deufel CL, Kavanaugh JA, Grams MP. Highs and Lows of Spatially Fractionated Radiation Therapy: Dosimetry and Clinical Outcomes. Pract Radiat Oncol. 2025 Jul-Aug;15(4):e388-e395. doi: 10.1016/j.prro.2024.12.002. Epub 2024 Dec 24. PMID 39725127
- [Background] Grams MP, Deufel CL, Kavanaugh JA, Corbin KS, Ahmed SK, Haddock MG, Lester SC, Ma DJ, Petersen IA, Finley RR, Lang KG, Spreiter SS, Park SS, Owen D. Clinical aspects of spatially fractionated radiation therapy treatments. Phys Med. 2023 Jul;111:102616. doi: 10.1016/j.ejmp.2023.102616. Epub 2023 Jun 11. PMID 37311338
- [Background] Crombe A, Kind M, Fadli D, Miceli M, Linck PA, Bianchi G, Sambri A, Spinnato P. Soft-tissue sarcoma in adults: Imaging appearances, pitfalls and diagnostic algorithms. Diagn Interv Imaging. 2023 May;104(5):207-220. doi: 10.1016/j.diii.2022.12.001. Epub 2022 Dec 23. PMID 36567193
- [Background] Oberoi S, Choy E, Chen YL, Scharschmidt T, Weiss AR. Trimodality Treatment of Extremity Soft Tissue Sarcoma: Where Do We Go Now? Curr Treat Options Oncol. 2023 Apr;24(4):300-326. doi: 10.1007/s11864-023-01059-2. Epub 2023 Mar 6. PMID 36877374
- [Background] Hoefkens F, Dehandschutter C, Somville J, Meijnders P, Van Gestel D. Soft tissue sarcoma of the extremities: pending questions on surgery and radiotherapy. Radiat Oncol. 2016 Oct 12;11(1):136. doi: 10.1186/s13014-016-0668-9. PMID 27733179
- [Background] Li H, Mayr NA, Griffin RJ, Zhang H, Pokhrel D, Grams M, Penagaricano J, Chang S, Spraker MB, Kavanaugh J, Lin L, Sheikh K, Mossahebi S, Simone CB, Roberge D, Snider JW, Sabouri P, Molineu A, Xiao Y, Benedict SH. Overview and Recommendations for Prospective Multi-institutional Spatially Fractionated Radiation Therapy Clinical Trials. Int J Radiat Oncol Biol Phys. 2024 Jul 1;119(3):737-749. doi: 10.1016/j.ijrobp.2023.12.013. Epub 2023 Dec 17. PMID 38110104
- [Background] O'Sullivan B, Davis AM, Turcotte R, Bell R, Catton C, Chabot P, Wunder J, Kandel R, Goddard K, Sadura A, Pater J, Zee B. Preoperative versus postoperative radiotherapy in soft-tissue sarcoma of the limbs: a randomised trial. Lancet. 2002 Jun 29;359(9325):2235-41. doi: 10.1016/S0140-6736(02)09292-9. PMID 12103287
- [Background] Spalato-Ceruso M, Ghazzi NE, Italiano A. New strategies in soft tissue sarcoma treatment. J Hematol Oncol. 2024 Sep 2;17(1):76. doi: 10.1186/s13045-024-01580-3. PMID 39218932
- [Background] Gamboa AC, Gronchi A, Cardona K. Soft-tissue sarcoma in adults: An update on the current state of histiotype-specific management in an era of personalized medicine. CA Cancer J Clin. 2020 May;70(3):200-229. doi: 10.3322/caac.21605. Epub 2020 Apr 10. PMID 32275330